CLINICAL TRIAL: NCT05378152
Title: Is Pipelle Biopsy of Benefit in Patients With Postmenopausal Bleeding and an Atrophic-appearing Cavity?
Brief Title: Assessing the Benefit of Pipelle Biopsy in Patients With Postmenopausal Bleeding and an Atrophic-appearing Cavity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: The Rotunda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: REC-2021-025
Record Dates: First submitted 2022-05-03; First posted 2022-05-18 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Postmenopausal Bleeding; Endometrial Cancer; Endometrial Hyperplasia
Keywords: Postmenopausal bleeding; Ambulatory gynaecology; Endometrial sampling; Endometrial hyperplasia; Endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pipelle biopsy (Active Comparator): This group will undergo an endometrial biopsy performed using a Pipelle catheter in the usual manner performed according to the physician either with or without a speculum and with or without a tenaculum. Local anaesthetic block may or may not be used as per clinical judgement.
  Interventions: Device: Pipelle biopsy catheter
- No Pipelle biopsy (Sham Comparator): This group will undergo a sham procedure where a speculum is inserted into the vagina and then removed.
  Interventions: Device: Sham procedure

INTERVENTIONS:
Device: Pipelle biopsy catheter — A speculum will be inserted into the vagina. A Pipelle biopsy catheter will be inserted through the cervix up to the fundus of the uterus. The internal piston will be withdrawn to create negative pressure. The catheter will be moved back and forth and rotated to collect the biopsy. The catheter will then be removed, followed by the speculum. The sample will be sent to the laboratory for assessment.
  Arms: Pipelle biopsy
Device: Sham procedure — A speculum is inserted into the vagina and then removed
  Arms: No Pipelle biopsy

SUMMARY:
Postmenopausal bleeding (PMB) is the occurrence of vaginal bleeding 12 months following a woman's last menstrual cycle. PMB represents one of the most common reasons for referral to gynaecology services. Approximately 10% of women with PMB will be found to have endometrial cancer. The gold standard of investigation of PMB is ambulatory gynaecology through the outpatient hysteroscopy clinic, which is often combined with Pipelle biopsy for endometrial sampling.

Up to 60% of women that present with PMB will have an atrophic-appearing cavity at hysteroscopy. This provides a challenge in obtaining a histological sample through both dilatation & curretage (D&C) and Pipelle biopsy. Often, scant tissue that is insufficient for clinical diagnosis is obtained.

Pipelle biopsy is associated with patient discomfort. It is also associated with costs related to the purchasing of equipment and the processing of samples in the laboratory to the sum of approximately 30 euro per sample. It is rare that a sample taken from an atrophic cavity will return any clinically meaningful result. A negative hysteroscopy reduces the probability of endometrial cancer to 0.6%.

This study aims to compare patients with PMB and atrophic-appearing cavity that undergo pipelle biopsy to those that do not. Differences in pain scores, cost saving and differences in clinical follow up will be assessed to evaluate the benefit of Pipelle biopsy in patients with PMB and atrophic-appearing cavity.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal
* Postmenopausal bleeding
* Tolerates hysteroscopy

Exclusion Criteria:

* Premenopausal
* Any lesion requiring biopsy at time of hysteroscopy
* Obvious cause of bleeding from the vagina or cervix at time of hysteroscopy
* History of endometrial hyperplasia/cancer

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-09-24 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
Pain scores | Immediately before procedure, less than 5 minutes prior to starting hysteroscopy
  Pain scores between groups using a 100mm visual analogue pain scale, with 100mm representing the highest level of pain
Pain scores | Immediately after procedure, within 1 minute of finishing hysteroscopy
  Pain scores between groups using a 100mm visual analogue pain scale, with 100mm representing the highest level of pain
Pain scores | Immediately after intervention, within 1 minute of carrying out intervention
  Pain scores between groups using a 100mm visual analogue pain scale, with 100mm representing the highest level of pain

SECONDARY OUTCOMES:
Cost saving | 3 months
  Cost saving between the two groups
Changes in follow up | 3 months
  Changes in follow up between groups including the number of repeat OPH assessments, follow up visits, repeat ultrasound scans and other related hospital attendances.,

CONTACTS AND LOCATIONS:
Locations (1):
- Rotunda hospital, Dublin, Ireland

REFERENCES:
- [Derived] Tunney DE, Yambasu DS, Gyawali DI, Gaughan DE, O'Dwyer DV, Harrity DC, Reidy DF, Ahmed DR, Molphy DZ, Asandei D, Salameh DF, Burke DN. Endometrial Biopsy Versus No Endometrial Biopsy with a Normal-Appearing Cavity During In-office Hysteroscopy for Postmenopausal Bleeding: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2025 Oct;32(10):914-920. doi: 10.1016/j.jmig.2025.07.007. Epub 2025 Jul 14. PMID 40669559